CLINICAL TRIAL: NCT00057551
Title: CBASP Augmentation for Treatment of Chronic Depression
Brief Title: Research Evaluating the Value of Augmenting Medication With Psychotherapy
Acronym: REVAMP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: U01MH062475 (NIH); U01MH062475 (NIH); U01MH061504 (NIH); U01MH061562 (NIH); U01MH061587 (NIH); U01MH061590 (NIH); U01MH062465 (NIH); U01MH062491 (NIH); U01MH062546 (NIH); U01MH063481 (NIH)
Record Dates: First submitted 2003-04-04; First posted 2003-04-07 (Estimated); Results first posted 2016-06-10 (Estimated); Last update posted 2017-12-06 (Actual); Status verified 2017-11

CONDITIONS: Depression; Depressive Disorder
MeSH Terms: conditions — Depression; Depressive Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBASP (Experimental): Cognitive Behavioral System of Psychotherapy plus medication (Could be switch to or addition of escitalopram, bupropion, venlafaxine or mirtazapine)
  Interventions: Behavioral: CBASP
- Brief Supportive Psychotherapy (Active Comparator): Brief Supportive Psychotherapy plus medication (Could be switch to or addition of escitalopram, bupropion, venlafaxine or mirtazapine)
  Interventions: Behavioral: Brief Supportive Psychotherapy
- Medication Only (Active Comparator): Could be switch to or addition of escitalopram, bupropion, venlafaxine or mirtazapine
  Interventions: Drug: Medication Only

INTERVENTIONS:
Behavioral: Brief Supportive Psychotherapy — brief supportive psychotherapy
  Arms: Brief Supportive Psychotherapy
Behavioral: CBASP — psychotherapy developed for chronic depression
  Other Names: Cognitive Behavioral Analysis System of Psychotherapy
  Arms: CBASP
Drug: Medication Only — antidepressant medication
  Other Names: one of five antidepressants
  Arms: Medication Only

SUMMARY:
This 24-week study, with a 12-month follow up period, will compare the effectiveness of antidepressant medication alone to the combination of psychotherapy and antidepressant medication in patients with chronic depression.

DETAILED DESCRIPTION:
Chronic depression affects approximately 5% of adults in the United States and is associated with significant functional impairment and high health care utilization. The combination of drug treatment and psychotherapy may be most effective in treating depression. This study will determine the effects of adjunctive psychotherapy in depressed patients who have failed to respond or have responded only partially to an initial trial medication.

Participants receive an initial trial of antidepressant medication for 8 to 12 weeks. Participants who continue to have depressive symptoms are randomly assigned to add Cognitive Behavioral Analysis System of Psychotherapy (CBASP) or supportive therapy to their medication regimens or to continue pharmacotherapy alone for an additional 12 weeks. Assessments are made at 6 and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria

* Major depressive episode
* Depressive symptoms > 2 years without remission
* Hamilton Depression Scale (HAM-D) score > 20
* Fluent in English

Exclusion Criteria

* Psychotic disorders, bipolar disorder, post traumatic stress disorder, obsessive compulsive disorder, or eating disorder
* Serious, unstable, or terminal medical condition
* Axis II diagnosis of antisocial, schizotypal, or severe borderline personality disorder
* Previous treatment with CBASP
* Previous ineffective treatment with 4 of the medication treatments used in the study
* Substance abuse
* Pregnancy
* Not willing to end other psychiatric treatment

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 491 (Actual)
Dates: Start 2003-04; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James H Kocsis, Principal Investigator — weill cornell mc
Locations (8):
- United States (8):
  - University of Arizona, Tucson, Arizona
  - Stanford University, Palo Alto, California
  - Emory University, Atlanta, Georgia
  - Weill-Cornell Medical College Payne Whitney Clinic, New York, New York
  - SUNY- Stony Brook, New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown University, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keller MB, McCullough JP, Klein DN, Arnow B, Dunner DL, Gelenberg AJ, Markowitz JC, Nemeroff CB, Russell JM, Thase ME, Trivedi MH, Zajecka J. A comparison of nefazodone, the cognitive behavioral-analysis system of psychotherapy, and their combination for the treatment of chronic depression. N Engl J Med. 2000 May 18;342(20):1462-70. doi: 10.1056/NEJM200005183422001. PMID 10816183
- [Background] Keller MB, Kocsis JH, Thase ME, Gelenberg AJ, Rush AJ, Koran L, Schatzberg A, Russell J, Hirschfeld R, Klein D, McCullough JP, Fawcett JA, Kornstein S, LaVange L, Harrison W. Maintenance phase efficacy of sertraline for chronic depression: a randomized controlled trial. JAMA. 1998 Nov 18;280(19):1665-72. doi: 10.1001/jama.280.19.1665. PMID 9831997
- [Background] McCullough JP Jr. Treatment for chronic depression using Cognitive Behavioral Analysis System of Psychotherapy (CBASP). J Clin Psychol. 2003 Aug;59(8):833-46. doi: 10.1002/jclp.10176. PMID 12858425
- [Derived] Shankman SA, Gorka SM, Katz AC, Klein DN, Markowitz JC, Arnow BA, Manber R, Rothbaum BO, Thase ME, Schatzberg AF, Keller MB, Trivedi MH, Kocsis JH. Side Effects to Antidepressant Treatment in Patients With Depression and Comorbid Panic Disorder. J Clin Psychiatry. 2017 Apr;78(4):433-440. doi: 10.4088/JCP.15m10370. PMID 28068460
- [Derived] Shankman SA, Campbell ML, Klein DN, Leon AC, Arnow BA, Manber R, Keller MB, Markowitz JC, Rothbaum BO, Thase ME, Kocsis JH. Dysfunctional attitudes as a moderator of pharmacotherapy and psychotherapy for chronic depression. J Psychiatr Res. 2013 Jan;47(1):113-21. doi: 10.1016/j.jpsychires.2012.09.018. Epub 2012 Oct 25. PMID 23102821
- [Derived] Klein DN, Leon AC, Li C, D'Zurilla TJ, Black SR, Vivian D, Dowling F, Arnow BA, Manber R, Markowitz JC, Kocsis JH. Social problem solving and depressive symptoms over time: a randomized clinical trial of cognitive-behavioral analysis system of psychotherapy, brief supportive psychotherapy, and pharmacotherapy. J Consult Clin Psychol. 2011 Jun;79(3):342-52. doi: 10.1037/a0023208. PMID 21500885
- [Derived] Kocsis JH, Gelenberg AJ, Rothbaum BO, Klein DN, Trivedi MH, Manber R, Keller MB, Leon AC, Wisniewski SR, Arnow BA, Markowitz JC, Thase ME; REVAMP Investigators. Cognitive behavioral analysis system of psychotherapy and brief supportive psychotherapy for augmentation of antidepressant nonresponse in chronic depression: the REVAMP Trial. Arch Gen Psychiatry. 2009 Nov;66(11):1178-88. doi: 10.1001/archgenpsychiatry.2009.144. PMID 19884606

RESULTS

PARTICIPANT FLOW:
Groups:
- CBASP: Cognitive Behavioral Analysis System of Psychotherapy
- BriefSP: Brief Supportive Psychotherapy
- Medication Only: An algorithm including Sertraline, Escitalopram
  Bupropion SR or XL
  Venlafaxine XR
  Mirtazapine
Period: Overall Study
Arm/Group | CBASP | BriefSP | Medication Only
Started | 200 | 195 | 96
Completed | 175 | 168 | 80
Not Completed | 25 | 27 | 16

BASELINE CHARACTERISTICS:
Groups:
- Brief Supportive P: Brief Supportive Psychotherapyherapy
- Medication Only: Sertraline
  Escitalopram
  Bupropion SR or XL
  Venlafaxine XR
  Mirtazapine
- Total: Total of all reporting groups
Arm/Group | CBASP | Brief Supportive P | Medication Only | Total
Number analyzed (Participants) | 200 | 195 | 96 | 491
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.2 (13.4) | 46.4 (11.7) | 45.3 (11.9) | 45.9 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 112 | 113 | 47 | 272
  Male | 88 | 82 | 49 | 219
Region of Enrollment [Number; unit: participants]
  United States | 200 | 195 | 96 | 491
Hamilton Depression Scale [Mean (Standard Deviation); unit: units on a scale] — Scores range from 0-72 with higher scores indicating more severe depression
  units on a scale | 19.52 (8.26) | 19.44 (8.31) | 18.4 (8.8) | 19.48 (8.27)

OUTCOME MEASURES:

1. Primary Outcome: Remission
Description: Hamilton Depression Scale (HAM-D)<8 and does not meet DSM-IV criteria for Major Depressive Disorder for 2 consecutive visits
Time Frame: 12 weeks
Population: Refers to # of subjects who completed 12 weeks of treatment
Measure: Number; unit: percentage of participants
Groups:
- Brief SP: Supportive Therapy
Arm/Group | CBASP | Brief SP | Medication Only
Number analyzed (Participants) | 174 | 168 | 76
percentage of participants | 38.5 | 31.0 | 39.5

ADVERSE EVENTS:
Groups:
- BriefSP: Supportive Therapy
- Medication: Sertraline
  Escitalopram
  Bupropion SR or XL
  Venlafaxine XR
  Mirtazapine
Arm/Group | CBASP | BriefSP | Medication
Serious Adverse Events (participants affected / at risk) | 0/200 | 0/195 | 0/96
Other Adverse Events (participants affected / at risk) | 28/200 | 23/195 | 8/96
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBASP (N=200) | BriefSP (N=195) | Medication (N=96)
moderate burden (Psychiatric disorders) | 28 (28) | 23 | 8 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No